CLINICAL TRIAL: NCT06306729
Title: Comparing the In-vivo Haemodynamic and Biomechanical Performance of Rapid-deployment Edwards Intuity Elite System and Edwards Magna Ease Valve
Brief Title: Computational Assessment of Bioprosthetic Aortic Valve Function
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Edwards Lifesciences (Industry); Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 316308
Record Dates: First submitted 2024-01-12; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: CFD; Valve Heart Disease
Keywords: Bioprosthesis
MeSH Terms: conditions — Heart Valve Diseases | interventions — Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Standard Implantation
  Interventions: Diagnostic Test: Computed Tomography, Magnetic Resonance Imaging
- Rapid Deployment
  Interventions: Diagnostic Test: Computed Tomography, Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Computed Tomography, Magnetic Resonance Imaging — Computed Tomography, Magnetic Resonance Imaging

SUMMARY:
Bioprosthetic valves are usually made of biological tissue that are mounted to a frame and are designed to function similarly to a healthy natural valve. Edwards Magna Ease and Intuity Elite bioprosthetic valves have similar leaflets and mounting designs. However, the valves are implanted in the patient in different ways (one is stitched to the wall of the left ventricular outflow tract, and the other is held in place by the radial force of the valve skirt). The study aims to understand in more detail how the different valves interact with the left ventricular outflow tract and aortic root.

DETAILED DESCRIPTION:
The implantation of a bioprosthetic valve is the established surgical technique when replacing the aortic valve to treat various aortic valve diseases. Many different bioprosthetic valves are available. The design and implantation technique in each system would result in different interaction with the left ventricular outflow tract (LVOT) and the aortic root, leading to different flow profiles that may induce platelet aggregation and affect the long-term performance of the bioprosthesis and its durability. Additionally, complications such as valve thrombosis may occur. However, it is not currently clear which bioprostheses/patients are more prone to thrombosis or degradation of the valve. This study aims to develop fluid-structure interaction (FSI) models, which can model blood flow and wall/valve mechanics, using realistic patient-specific geometries and flow conditions which correlate with the true performance of the valve in the imaged patients, and to assess and compare such performances to understand the benefits and challenges with various bioprosthetic valves.

FSI models combine computational fluid mechanics (CFD) with structural wall mechanics modelling. This is an alternative approach that allows detailed assessment of flow patterns and estimation of wall shear stress and pressure within blood vessels, and therefore has been applied increasingly to gain better insights into the hemodynamics in cardiovascular diseases

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years or over.
* Patients diagnosed with aortic valve disease, and scheduled to undergo Edwards Magna Ease or Intuity Elite and free of exclusion criteria below.
* The patient is willing and able to understand the Patient Information Sheet and provide written informed consent.
* The patient must agree to comply with the study imaging protocol as required at prespecified times.

Exclusion Criteria:

* Inability to provide valid informed consent.
* Male and female patients aged < 18 years of age.
* Contraindications for CT angiography: renal failure (Cr>250 μmol/L or eGFR<30 mL/min) due to the additional risk of contrast medium nephrotoxicity or allergy to iodine.
* Women of childbearing age who have not had a hysterectomy and/or who may be breastfeeding.
* History of cardiac pacing device insertion, or any other MRI incompatible device implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 informed and consented patients who undergo the Intuity Elite (n=10) and Magna EASE (n=10) valves will be prospectively enrolled. The patients will be evaluated at 3- and 12-months post valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
blood flow velocities | 12 months
  Blood flow velocities (cm/s) will be quantified for each bioprosthesis at 3 levels: subvalvular (LVOT and native annulus), transvalvular, the aortic root, and the proximal ascending aorta. Velocities more than 20cm/s will be taken as abnormal.
Time average wall shear stress (TAWSS) | 12 months
  TAWSS will be quantified for each bioprosthesis at 3 levels: subvalvular (LVOT, the aortic root, and the proximal ascending aorta. TAWSS under 0.5Pa is taken as low, 0.51-2.0 as moderately increased, >2.0 Pa as severely increased TAWSS.

SECONDARY OUTCOMES:
Patient's satisfaction | 12 months
  A questionnaire will be designed to score valve-related clinical symptoms following the intervention.
Evidence of major adverse cardiac and cerebrovascular events (MACCE) | 12 months
  Evidence of MACCE (Stroke and myocardial infarction in the first 12 months post procedure)
Mortality | 12 months
  Evidence of mortality during the 12 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Mirsadraee, MD, Ph.D, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No